CLINICAL TRIAL: NCT02766803
Title: Prospective, Randomized, Double - Blind Placebo Controlled Trial of Simvastatin and Resveratrol Therapy on Clinical, Endocrinological, Biochemical and Endothelial Dysfunction Parameters in Women With Polycystic Ovary Syndrome.
Brief Title: Effects of Simvastatin and Micronized Trans-resveratrol Treatment on Polycystic Ovary Syndrome (PCOS) Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Beata Banaszewska, MD PhD Ass Professor, Poznan University of Medical Sciences
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PoznanUMS 3
Record Dates: First submitted 2016-05-09; First posted 2016-05-10 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: PCOS, Insulin Resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin + resveratrol (Active Comparator): simvastatin 20 mg daily micronized trans-resveratrol 500 mg daily
  Interventions: Drug: Simvastatin and micronized trans-resveratrol
- simvastatin+ placebo (Placebo Comparator): simvastatin 20 mg daily Placebo
  Interventions: Drug: Simvastatin and micronized trans-resveratrol

INTERVENTIONS:
Drug: Simvastatin and micronized trans-resveratrol

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrinopathy affecting women of reproductive age. Hyperandrogenism is the central feature of PCOS. Studies on isolated ovarian theca-interstitial cells indicate that resveratrol, a natural polyphenol, reduces androgen production.

This study is designed to evaluate the endocrine and metabolic effects of simvastatin and resveratrol on PCOS.

Methods: A randomized (1:1) double-blind, placebo-controlled trial will evaluate the effects of administering 20 mg of simvastatin daily and 500 mg of resveratrol daily, or administering 20 mg simvastatin and the placebo to women with PCOS at an academic hospital. PCOS is defined according to the Rotterdam criteria. Evaluations are performed at baseline and repeated after 3 and 6 months of treatment. The main outcome is a change of the serum total testosterone and the fasting insulin level.

ELIGIBILITY:
Inclusion Criteria:

* PCOs
* insulin resistance
* normal prolactin, TSH, 17 OH progesterone No evidence of androgen producing malignancy, Cushing's syndrome or acromegaly

Exclusion Criteria:

* use of oral contraceptives and/or other steroid hormones 3 months prior to the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
testosterone serum concentration | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Infertility and Reproductive Endocrinology, Department of Gynecology and Obsterics, Poznan, Poland

REFERENCES:
- [Derived] Xiong T, Fraison E, Kolibianaki E, Costello MF, Venetis C, Kostova EB. Statins for women with polycystic ovary syndrome not actively trying to conceive. Cochrane Database Syst Rev. 2023 Jul 18;7(7):CD008565. doi: 10.1002/14651858.CD008565.pub3. PMID 37462232